CLINICAL TRIAL: NCT06431802
Title: Construction and Application of the Visualization Training Platform Based on a Multimodal Standardized Dataset for Pain Assessment in Critically Ill Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FNF20231219
Record Dates: First submitted 2024-05-17; First posted 2024-05-29 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Pediatrics; Critical Illness; Pain Measurement
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional intervention group (Active Comparator): On-site course training in pain assessment
  Interventions: Other: Conventional intervention
- Platform intervention group (Experimental): Pain assessment training using the visualization training platform based on a multimodal standardized dataset for pain assessment in critically ill children
  Interventions: Behavioral: Platform intervention

INTERVENTIONS:
Other: Conventional intervention — A nursing specialist with extensive clinical and teaching experience will provide on-site course training. The training will cover topics related to pain and pain assessment, such as: pain definition, types, physiological mechanisms, performance, pain assessment tools, and frequency of pain assessment. Interventions will be provided once a week for 4 weeks.
  Arms: Conventional intervention group
Behavioral: Platform intervention — Using a pre-assigned account to log in to the platform, read the guidance instructions and enter the platform to start training. Basic knowledge of pain and pain assessment can be learnt through the Learning Resources module on the platform, and pain assessment training can be conducted through the Pain Assessment Exercise module. During pain assessment training the platform provides instant feedback based on the participant's exercises. Interventions will be completed in 4 weeks.
  Arms: Platform intervention group

SUMMARY:
The goal of this clinical trial is to learn if the visualization training platform based on a multimodal standardized dataset for pain assessment in critically ill children is applicable for pain assessment training. The study aims to answer:

1. Does pain assessment training with a visualization training platform based on a multimodal standardized dataset for pain assessment in critically ill children improve participants' knowledge level of pain assessment?
2. Does pain assessment training with a visualization training platform based on a multimodal standardized dataset for pain assessment in critically ill children improve participants' skill level of pain assessment?

Researchers will compare a visualization training platform based on a multimodal standardized dataset for pain assessment in critically ill children to on-site lessons to see how well the platform intervention can be applied to pain assessment training.

Participants will:

1. Use the visualization platform or receive on-site lessons for pain assessment training every week for 1 month.
2. Test before and 1 month after the start of the study.

DETAILED DESCRIPTION:
In pediatric intensive care units, children are often faced with complex and critical conditions that require frequent procedures which may cause pain, and experience varying degrees of pain. Pain can have serious negative effects on the physiological, psychological, and social well-being of critically ill children, and may even lead to long-term distress, impeding both individual growth and overall health. Reliable pain assessment can help healthcare professionals to better understand the type and extent of pain in children, so that appropriate interventions can be taken to better manage the child's pain and thereby improve the child's health outcomes. However, pediatric nurses face challenges from the child, observational indicators, and the individual themselves during pain assessment in the clinic. Training in pain assessment can effectively improve nurses' knowledge, skills and attitudes, enabling them to better cope with the difficulties associated with pain assessment, thereby improving the quality of pain management and providing optimal pain care for children. Traditional training has many drawbacks, and there are various difficulties in pain assessment training for critically ill children, which brings various challenges to pain assessment training for pediatric ICU nurses. Visualization training, being intuitive, interactive, and personalized, offers unique advantages over traditional training methods. The union of deliberate practice with visualization training can further enhance the training effect, and help pediatric ICU nurses' pain assessment ability to be comprehensively improved through purposeful practice, timely feedback, and repeated training and challenges, so that they can more accurately identify and assess children's pain. Therefore, a visualization training platform based on a multimodal standardized dataset for pain assessment in critically ill children will be constructed for pain assessment training to promote better improvement of pain assessment ability of pediatric ICU nurses, so that pain in critically ill children can be better managed.

ELIGIBILITY:
Inclusion Criteria:

1. Obtain a Nurse Practitioner's Certificate;
2. Nurses working in critical care;
3. Voluntarily participate in this study.

Exclusion Criteria:

1. Nurses in the neonatal unit (due to the specificity of pain assessment in neonates);
2. Not on duty during the survey period due to further training, rotations, sick leave, maternity leave, etc.;
3. Nurses who travel to our hospital for further training, rotations, or clinical placements during the survey period;
4. Those who fail to complete the full intervention or withdrew from the study midway.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Knowledge level of pain assessment | baseline, 1st month since baseline
  Use the Pediatric ICU Nurses' Pain Assessment Knowledge Test，which is measured on a scale from 0 to 100 points. The higher the total score, the higher the level of knowledge.
Skill level of pain assessment | baseline, 1st month since baseline
  The pediatric pain assessment cases developed by the research team will be utilized for evaluation. The correct percentage range is from 0% to 100%, with higher percentages indicating a higher skill level in pain assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Gu, Doctor, Study Director — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China